CLINICAL TRIAL: NCT01447381
Title: Systemic Therapies for Pediatric Atopic Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rady Children's Hospital, San Diego (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Wynnis Tom, MD, Assistant Clinical Professor, Rady Children's Hospital, San Diego
Other Study IDs: CMH 2011-14488
Record Dates: First submitted 2011-08-11; First posted 2011-10-06 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- mycophenolate mofetil: Moderate to severe atopic dermatitis being treated with systemic mycophenolate mofetil
- cyclosporine: Moderate to severe atopic dermatitis being treated with systemic cyclosporine
- azathioprine: Moderate to severe atopic dermatitis being treated with systemic azathioprine
- methotrexate: Moderate to severe atopic dermatitis being treated with systemic methotrexate

SUMMARY:
While many patients with atopic dermatitis (eczema) can be managed with topical creams and treatments for itch, some children have such severe, long-standing disease that they need treatment with oral medications that decrease the ability of the immune system to react. However, there is not enough information on the proper use of these medications or how well they work compared with each other. The current study looks at the response of children treated with these medications to provide this information and improve their use.

DETAILED DESCRIPTION:
Severe and/or refractory cases of atopic dermatitis (AD) can require systemic immunosuppressive therapy for disease control, yet there are few studies regarding the appropriate use of these drugs for pediatric AD and even less data comparing them. The current observational study will observe the effect of these therapies on children with moderate to severe atopic dermatitis as they are treated. These drugs being observed will be cyclosporine, azathioprine, mycophenolate mofetil, and methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate, severe, or very severe atopic dermatitis meeting the Hanifin and Rajka criteria
* Needs systemic therapy (e.g. cyclosporine, azathioprine, mycophenolate mofetil, or methotrexate) for severe atopic dermatitis
* Subject has severe or recalcitrant disease interrupting daily life as evidenced by fulfilling 2 or more of the following 4 criteria:

  * Failure of multimodal therapy including emollients/barrier repair, topical anti-inflammatory agents (medium to high potency topical corticosteroids, and/or low-potency or topical calcineurin inhibitors if facial/intertriginous areas), and antihistamines
  * Significant impairment in quality of life (physical, psychological, emotional) such as significant sleep disruption, poor school performance, or frequent school absenteeism, per the judgement of the investigator.
  * Inability to receive, prior failure, or the need for more than one course of phototherapy
  * Prior failure or need for more than one course of another oral immunosuppressive medication
* No serious medical condition that precludes the use of oral immunosuppressives based on the subject's medical history, physical examination, and safety laboratory tests.
* Negative PPD within the last year prior to study initiation.
* Female of childbearing potential has a negative pregnancy test at the time of starting the systemic drug and who consents to be abstinent or using an effective method of contraception during the study. Effective contraception is defined as IUD, condom with spermicide, diaphragm with spermicide, or stable use of a hormonal contraceptive (oral, implant, injection or transdermal patch) beginning at least 1 month prior to starting the systemic drug.
* Subject and parent/guardian are willing and able to comply with study instructions and return to the clinic for all required visits.

Exclusion Criteria:

* Female who is pregnant, nursing, or planning a pregnancy during the study period.
* Concurrent participation in another clinical trial with an investigational drug or device that may impact on the individual's atopic dermatitis.
* Subjects with clinically significant hepatic disease, history of lymphoma or myelosuppression, low TMPT activity (if starting azathioprine), renal disease (if starting cyclosporine or azathioprine), hypertension (if starting cyclosporine), blood dyscrasias, or central nervous system disorders, such as uncontrolled seizures or peripheral neuropathy, or taking systemic medications that could interact adversely with the study medicine (e.g. erythromycin use with cyclosporine).
* Subjects with any underlying disease that the Investigator deems uncontrolled, and poses a concern for subject safety while participating on the study.
* Subject has a history of clinically significant drug or alcohol abuse in the last year.
* Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
* Active systemic infection that could worsen with systemic therapy for AD.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Ages 2 to 17 (inclusive) with moderate to severe atopic dermatitis and who require treatment with cyclosporine, azathioprine, mycophenolate mofetil, and/or methotrexate. Both male and female. Non-pregnant females and minorities will be included without restriction.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2011-10; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in Investigator Global Severity Scale (IGSS) | 10 years
Reduction in SCORing Atopic Dermatitis (SCORAD) Index | 10 years
Reduction in Eczema Area and Severity Index (EASI) | 10 years

SECONDARY OUTCOMES:
Time to Response | 10 years
Rate of Taper | 10 years
  Measuring the rate of dose descalation of systemic immunosuppresive without increase in atopic dermatitis severity as measured by IGSS, SCORAD and EASI assessments.
Length of time before recurrent flare | 10 years
  Durability of response is the measure of time before recurrent flare after discontinuation of systemic immunosuppressive therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wynnis Tom, MD, Principal Investigator — Rady Children's Hospital and UC San Diego
Locations (3):
- United States (3):
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's Memorial Hospital, Chicago, Illinois

REFERENCES:
- [Background] Meagher LJ, Wines NY, Cooper AJ. Atopic dermatitis: review of immunopathogenesis and advances in immunosuppressive therapy. Australas J Dermatol. 2002 Nov;43(4):247-54. doi: 10.1046/j.1440-0960.2002.00610.x. PMID 12423430
- [Background] Akhavan A, Rudikoff D. The treatment of atopic dermatitis with systemic immunosuppressive agents. Clin Dermatol. 2003 May-Jun;21(3):225-40. doi: 10.1016/s0738-081x(02)00362-0. No abstract available. PMID 12781440